CLINICAL TRIAL: NCT07098286
Title: Enhancing Resilience Among Patients With Stroke: Implementation of High Intensity Home-based Rehabilitation
Acronym: HIHR
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Claude D. Pepper Older American Independence Centers (OAICS) (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00114972
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Stroke Rehabilitation
Keywords: Rehabilitation Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- High intensity home-based rehabilitation (HIHR) prospective cohort at Duke: The HIHR cohort at Duke will be the prospective intervention cohort. They will receive occupational, physical, and speech therapy services at frequencies that are greater than standard home care after a stroke. They may also receive home health aide services if deemed clinically appropriate. Data for this cohort of patients will be combined with data from the HIHR cohort at Cleveland Clinic and will be compared to data from the inpatient rehabilitation facility (usual care) retrospective cohort. These patients will also participate in phone-based surveys and may also choose to participate (with their primary at-home caregiver) in an interview with a study team member.
  Interventions: Other: high intensity home-based rehabilitation
- Inpatient rehabilitation facility (usual care) retrospective cohort: These patients' data will be accessed retrospectively using the electronic health record at both Duke and Cleveland Clinic, and a Medicare database. Their data will be included if their hospital data confirms that they were eligible for discharge to HIHR but were discharged to an inpatient rehabilitation facility for post-acute rehabilitation. Data will be included if the hospital discharge occurred between October 2021 and December 2024. Data for this cohort of patients will be compared to data from the HIHR cohorts at both Duke and Cleveland Clinic.
- High intensity home-based rehabilitation (HIHR) retrospective cohort at Cleveland Clinic: This will be a retrospectively identified cohort of patients who were admitted to a Cleveland Clinic hospital for treatment of a stroke then discharged home to receive HIHR services from Cleveland Clinic Home Care. Data will be included for patients if their HIHR episode occurred between October 2021 and December 2024. Data for this cohort of patients will be combined with data from the HIHR cohort at Duke and will be compared to data from the inpatient rehabilitation facility (usual care) retrospective cohort.
- Inpatient rehabilitation facility (usual care) cohort at Duke: These will be patients admitted to Duke Hospital between August 2025 and July 2026 who met eligibility to discharge to HIHR but instead discharged to an inpatient rehabilitation facility. These patients will be contacted for potential study enrollment 30-60 days after their hospital discharge. If they consent to participate, they will respond to phone-based surveys with a member of the study team. They may also choose to participate (with their primary at-home caregiver) in an interview with a member of the study team.

INTERVENTIONS:
Other: high intensity home-based rehabilitation — Whereas standard home healthcare would include 1-3 visits per week of therapy services after a stroke, the HIHR intervention will include at least therapy visits per week. Between occupational, physical, and speech therapy, the frequency for each will match individual patient needs based on the type and severity of their stroke-related deficits.
  Groups: High intensity home-based rehabilitation (HIHR) prospective cohort at Duke

SUMMARY:
The goal of this observational study is to test whether a model of high-intensity home-based rehabilitation (HIHR) helps patients get good outcomes after treatment for a stroke at Duke University Hospital. The main question it aims to answer is:

Do patients who receive HIHR services after their stroke recover their function at least as well as patients who discharge to an inpatient rehabilitation facility?

Participants will not be assigned to any group. Rather, patients who choose to discharge from the hospital to their home and receive HIHR services after their stroke will be enrolled in the study so that researchers can compare their outcomes to those for other patients who instead discharged to an inpatient rehabilitation facility.

DETAILED DESCRIPTION:
This study will test whether a model of high-intensity home-based rehabilitation (HIHR) helps patients get good outcomes after treatment for a stroke at Duke University Hospital. While research data for this study is being collected exclusively at Duke, it will be combined with data from Cleveland Clinic, where HIHR was developed and where patients can select it as a standard-of-care option for rehabilitation after their stroke. Data from patients in both hospital systems (i.e., a prospective HIHR cohort from Duke and a retrospective HIHR cohort from Cleveland Clinic) will be used to understand if patients' outcomes are at least as good when they use HIHR services compared to an inpatient rehabilitation facility. Researchers will use retrospective data from the Centers for Medicare and Medicaid services to compare outcomes for patients in the two HIHR cohorts to outcomes for similar patients in an inpatient rehabilitation facility cohort.

To study both the ability of clinicians to implement HIHR and the outcomes that patients achieve, no one will be assigned to HIHR as a participant in this study at Duke. Rather, during their hospitalization, patients who are being treated for a stroke can decide whether they are interested in using HIHR services when they discharge. Those who do will be enrolled in the study, becoming part of the HIHR cohort. They will discharge to their own home to receive HIHR services in their home. These services will include occupational, physical, and/or speech therapy for at least six hours per week, which is significantly more than patients normally receive when discharging home. If considered necessary, patients who choose HIHR and enroll in the study may also receive nursing care and up to 32 hours of services from a home health aide. The clinical team taking care of participants in HIHR will meet weekly to discuss progress and ongoing care plans. The HIHR care episode is expected to last approximately 14 days for each patient.

As follow-up for the study, every patient in the HIHR will be asked to respond to phone-based surveys with a member of the research team after their HIHR services end. Those who are interested can also participate in a 45-60 minute interview with one of the researchers. For those interviews, the patient's primary at-home caregiver will also be asked to enroll in the study in order to participate in the interview and share their experiences.

Separately, the research team will recruit via phone some patients who discharged from Duke Hospital to an inpatient rehabilitation facility after treatment for their stroke. Patients in that group who agree to participate will also complete the phone-based surveys and can participate (with their primary at-home caregiver) in an interview with one of the researchers. The survey responses and the interviews for the HIHR group and the group of patients discharged to rehabilitation facilities will be compared by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand English.
* Admitted to Duke University Hospital stroke medical service
* Confirmed diagnosis of stroke (per documentation in medical record)
* At time of hospital discharge:

  a) Home address in Durham County b) NIH Stroke Scale Score = 4-13 c) AM-PAC 6-Clicks basic mobility score >/=13 d) Documented need for post-acute rehabilitation from 2 disciplines e) No contraindications to safe medical management at home (ongoing cancer treatment, dialysis-dependent ESRD, complex wounds, others as determined by the attending medical team) g) Clinically judged to have adequate caregiver support at home

Exclusion Criteria:

* Those with acute psychosis or an inability to provide legal and effective consent will be excluded from participation.
* Those with medical contraindications as determined by the hospital attending neurology team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for an acute stroke at Duke University Hospital who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical function | From enrollment to the end of the HIHR episode, approximately 7-14 days.
  The primary outcome will be physical function as measured by the Continuity Assessment Record and Evaluation (CARE) section GG form. This form, required by CMS for all post-acute care settings, will provide separate scores reporting physical function domains of mobility and self-care. Scores for the mobility domain range from 15 to 90. Scores for the self-care domain range from 8 to 48. For both, higher scores indicate greater independence with tasks consistent with that domain (e.g., walking for the mobility domain and dressing for the self-care domain).

SECONDARY OUTCOMES:
Hospital length of stay | From enrollment to hospital discharge, expected 1-5 days
  Researchers will examine whether hospital length of stay is reduced when patients are able to discharge to HIHR.

OTHER OUTCOMES:
Self-reported physical function | Approximately 30-45 days after discharge from the hospital.
  Patients in both the HIHR and inpatient rehabilitation facility cohorts at Duke will respond to questions from the Patient Reported Outcome Measure Information System (PROMIS) physical function questionnaire. The computer-adapted version of this questionnaire will be used, meaning that patients will respond to 4-8 total questions. Researchers will use the PROMIS T-scale scores for this study. Those scores range from 0-100 with higher scores indicating higher levels of function.
Self-reported satisfaction with social roles | Approximately 30-45 days after discharge from the hospital
  Patients in both the HIHR and inpatient rehabilitation facility cohorts at Duke will respond to questions from the Patient Reported Outcome Measure Information System (PROMIS) satisfaction with social roles questionnaire. The computer-adapted version of this questionnaire will be used, meaning that patients will respond to 4-8 total questions. Researchers will use the PROMIS T-scale scores for this study. Those scores range from 0-100 with higher scores indicating higher levels of satisfaction with social roles.
Self-reported resilience | Approximately 30-45 days after hospital discharge
  Patients in both the HIHR and inpatient rehabilitation facility cohorts at Duke will respond to questions from the Brief Resilience Score questionnaire. The Brief Resilience Scale (BRS) is a validated self-report instrument designed to assess an individual's ability to recover from stress and adversity. It consists of six items rated on a 5-point Likert scale, with higher scores indicating greater resilience.
Perceived acceptability of HIHR as a model for post-stroke rehabilitation | Approximately 45-60 days after hospital discharge
  The subgroup of patients in the HIHR cohort at Duke who participate in the interviews will complete the Acceptability of Intervention Measure (AIM) in relation to the perception about HIHR as a model for post-stroke rehabilitation. The AIM includes 4 items, each with a 5-point Likert response. Total scores are 5-20 with higher scores indicating greater acceptability.
Perceived appropriateness of HIHR as a model for post-stroke rehabilitation | Approximately 45-60 days after hospital discharge
  The subgroup of patients in the HIHR cohort at Duke who participate in the interviews will complete the Intervention Appropriateness Measure (IAM) in relation to the perception about HIHR as a model for post-stroke rehabilitation. The IAM includes 4 items, each with a 5-point Likert response. Total scores are 5-20 with higher scores indicating greater perceived appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua K. Johnson, DPT, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No